CLINICAL TRIAL: NCT02514564
Title: The Effects of Aerobic Exercise Training in Patients With Cardiovascular Diseases Related to Microvascular Endothelium Function, Angiogenesis, Oxidative Stress and Aerobic Capacity
Brief Title: The Effects of Aerobic Exercise in Microvascular Endothelium Function in Patients With Cardiovascular Diseases
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Cardiologia de Laranjeiras (Other)
Responsible Party: Principal Investigator, Juliana Pereira Borges, PhD, Instituto Nacional de Cardiologia de Laranjeiras
Other Study IDs: Faperj-E-26/101.575
Record Dates: First submitted 2015-07-30; First posted 2015-08-03 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for nitrite/nitrate quantification.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 2x/wk: This group will be consisted of patients that will perform exercise two times a week.
  Interventions: Behavioral: Exercise
- 3x/wk: This group will be consisted of patients that will perform exercise three times a week.
  Interventions: Behavioral: Exercise
- Control: This group will not perform exercise.

INTERVENTIONS:
Behavioral: Exercise — Patients included in the study will be enrolled in a cardiac rehabilitation program, in an independent manner of the study protocols.
  Groups: 2x/wk; 3x/wk

SUMMARY:
This study evaluates the effects of different volumes of aerobic exercise training in cardiovascular parameters of patients with cardiovascular diseases enrolled in a cardiac rehabilitation program.

DETAILED DESCRIPTION:
Aerobic exercise training is well known to improve endothelium dependent vasodilatation in the microcirculation. However, the impact of exercise frequency on this response in patients with coronary artery disease remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* sedentarism for at least 6 months;
* clinical diagnosis for coronary artery disease (occurrence of any acute coronary syndrome, including ST elevation or non-ST elevation myocardial infarction or unstable angina or by the diagnosis of obstructive coronary artery disease on coronary angiography in patients with stable angina).

Exclusion Criteria:

* nephropathies;
* decompensated cardiovascular diseases;
* liver diseases.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in the hospital in which the exercise will be performed.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Changes in Skin microvascular blood flow | Change from baseline in skin microvascular blood flow at 6 months
  Measured through a Laser Speckle Contrast Imaging equipment

SECONDARY OUTCOMES:
Change in peak oxygen consumption | Change from baseline in peak oxygen consumption at 6 months
  Measured at a maximal graded exercise test
Change in weight | Change from baseline in weight at 6 months
  Measured with a calibrated digital scale

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo V Tibiriçá, PhD, Study Director — Instituto Fernandes Figueira
Locations (1):
- Instituto Nacional de Cardiologia, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Souza EG, De Lorenzo A, Huguenin G, Oliveira GM, Tibirica E. Impairment of systemic microvascular endothelial and smooth muscle function in individuals with early-onset coronary artery disease: studies with laser speckle contrast imaging. Coron Artery Dis. 2014 Jan;25(1):23-8. doi: 10.1097/MCA.0000000000000055. PMID 24172594
- [Background] Cordovil I, Huguenin G, Rosa G, Bello A, Kohler O, de Moraes R, Tibirica E. Evaluation of systemic microvascular endothelial function using laser speckle contrast imaging. Microvasc Res. 2012 May;83(3):376-9. doi: 10.1016/j.mvr.2012.01.004. Epub 2012 Jan 31. PMID 22326551
- [Derived] Borges JP, Mediano MF, Farinatti P, Coelho MP, Nascimento PM, Lopes GO, Kopiler DA, Tibirica E. The Effects of Unsupervised Home-based Exercise Upon Functional Capacity After 6 Months of Discharge From Cardiac Rehabilitation: A Retrospective Observational Study. J Phys Act Health. 2016 Nov;13(11):1230-1235. doi: 10.1123/jpah.2016-0058. Epub 2016 Aug 24. PMID 27333938